CLINICAL TRIAL: NCT07205848
Title: Evaluating Public Awareness and Preventive Actions for Dengue Fever in Sudan Amidst Ongoing Crises: A Community Survey on Knowledge and Practices in Line With Related SDGs
Brief Title: Evaluating Public Awareness and Preventive Actions for Dengue Fever in Sudan Amidst Ongoing Crises
Status: Completed | Type: Observational
Sponsor: Research and Publication office (Other)
Responsible Party: Sponsor
Other Study IDs: 24009
Record Dates: First submitted 2025-02-10; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2024-12

CONDITIONS: Dengue Hemorrhagic Fever; Awareness
Keywords: Dengue Fever; Sudan; Awareness; Prevention; Public
MeSH Terms: conditions — Severe Dengue; Dengue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sudanese nationals with internet access: Sudanese nationals with internet access
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study evaluates the awareness of dengue fever and preventive measures among Sudanese people during the war. It assesses knowledge, awareness, implementation of prevention, access to healthcare, community involvement, and the link between knowledge and practice. The findings aim to enhance disease control strategies in conflict settings.

DETAILED DESCRIPTION:
This study aims to evaluate the level of awareness of dengue fever and preventive measures among the Sudanese population during the war. The research focuses on understanding public knowledge, awareness, and the implementation of preventive actions in a conflict setting, aligning with various Sustainable Development Goals (SDGs).

The specific objectives include:

1. Measuring the knowledge level of the Sudanese population regarding dengue fever during the war (SDG 3, 4).
2. Evaluating awareness of preventive measures against dengue fever (SDG 3, 6).
3. Assessing the extent to which preventive measures are implemented (SDG 3, 11).
4. Investigating access to healthcare facilities during the dengue fever outbreak (SDG 3, 10).
5. Identifying the role of community participation in controlling the outbreak (SDG 3, 17).
6. Examining the correlation between knowledge levels and the implementation of preventive measures (SDG 3).

By addressing these objectives, the study aims to provide insights into public health challenges and community responses during the war, contributing to improved disease control strategies in conflict-affected areas

ELIGIBILITY:
- Inclusion Criteria: Sudanese nationals with internet access Residents in any part of Sudan age above or equal 17 years Individuals willing to participate

- Exclusion Criteria: Non Sudanese nationals. Sudanese nationals with no internet access Residence outside Sudan age less than 17 years

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sudanese individuals above or equal 17 years and above residing in any part of
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: Level of Knowledge: Percentage of the Sudanese population aware of dengue fever and its symptoms during the war | 1_2 months
  Using a structured, self-administered questionnaire (SAQ) based on a validated KAP survey on dengue fever.

SECONDARY OUTCOMES:
To measure the preventive knowledge against dengue fever | Jan - Mar 2025
  Using a structured, self-administered questionnaire (SAQ) based on a validated KAP survey on dengue fever, in the form of (True, False, I don't know) responses.
to measure the extent of implementation of preventive measures. | 1- 2 months
  Using a structured, self-administered questionnaire (SAQ) based on a validated KAP survey on dengue fever, in the form of Likert's scale responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Research and publication office, Khartoum, Omdurman, Sudan

IPD SHARING:
Plan to Share IPD: No